CLINICAL TRIAL: NCT07082387
Title: External Oblique and Rectus Abdominis Plane (EXORA) Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: External Oblique and Rectus Abdominis Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1261/6/25
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: External Oblique and Rectus Abdominis Plane Block; Quadratus Lumborum Block; Postoperative Analgesia; Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXORA group (Experimental): Patients will receive an external oblique and rectus abdominis plane (EXORA) block using 20ml of bupivacaine 0.25%.
  Interventions: Other: External oblique and rectus abdominis plane block
- QLB group (Experimental): Patients will receive a quadratus lumborum block (QLB) using 20ml of bupivacaine 0.25%.
  Interventions: Other: Quadratus lumborum block

INTERVENTIONS:
Other: External oblique and rectus abdominis plane block — Patients will receive an external oblique and rectus abdominis plane (EXORA) block using 20ml of bupivacaine 0.25%.
  Arms: EXORA group
Other: Quadratus lumborum block — Patients will receive a quadratus lumborum block (QLB) using 20ml of bupivacaine 0.25%.
  Arms: QLB group

SUMMARY:
This study aims to compare the effects of the external oblique and rectus abdominis plane (EXORA) block and the quadratus lumborum block (QLB) on postoperative analgesia in patients undergoing laparoscopic cholecystectomy (LC).

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is a proven, gold standard surgical procedure for the management of gallbladder stones.

The quadratus lumborum block (QLB) is a regional block that would appear to be similar to the posterior TAP block, although the drug injection area is deeper and more dorsal than the transverse abdominal aponeurosis.

The external oblique and rectus abdominis plane (EXORA) block is an emerging technique providing a sensory block to the anterolateral abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Undergoing laparoscopic cholecystectomy (LC) under general anesthesia.

Exclusion Criteria:

* History of allergies to local anesthetics.
* Opioid dependency.
* Bleeding or coagulation disorders.
* Psychiatric and neurological disorder.
* Local infection at the site of injection.
* Body mass index (BMI) > 35.
* Hypertension.
* Uncontrolled diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to first dose of morphine administrated).

SECONDARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4.
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 0.5 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at PACU, 2, 4, 6, 8, 12, 18 and 24 h postoperatively.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, pruritus, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.